CLINICAL TRIAL: NCT03928860
Title: The Effect of One Session Osteopathic Manuel Treatment on Femoral Artery Diameter and Flow in Patients With Peripheral Arterial Disease
Brief Title: The Effect of One Session Osteopathic Manuel Treatment on Femoral Artery Diameter and Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Muhammet Ayhan ORAL, Research Assistant, Kırıkkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAD AND ONE SESSION OMT
Record Dates: First submitted 2019-04-22; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral arterial disease; Osteopathic manual treatment
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OMT Session and Doppler Ultrasonography (Experimental): OMT Session Patients with PAD will be received 30 minutes of osteopathic manual treatment for one session. During application, the patient was in the supine position. OMT treatment session include, sub occipital release technique, supraclavicular release technique, sternal mobilization, omentum minus release, liver pumping, diaphragmatic mobilization, grand manevra technique, hip mobilization, knee mobilization and ankle mobilization. Each technique was applied for 3 minutes to patients.
  Doppler Ultrasonography Femoral artery diameter and flow evaluated by radiologist.
  In the evaluation, the wall contour characteristics of the vessel to be examined were evaluated and the diameter was measured. Color doppler examination was performed to determine whether the vessel contained color filling, patency, flow direction and turbulence.
  Peak systolic and end diastolic flow rates and flow pattern and flow rate were measured by spectral examination
  Interventions: Other: OMT session

INTERVENTIONS:
Other: OMT session — Patients with PAD will be received 30 minutes of osteopathic manual treatment for one session. During application, the patient was in the supine position. OMT treatment session include, sub occipital release technique, supraclavicular release technique, sternal mobilization, omentum minus release, liver pumping, diaphragmatic mobilization, grand manevra technique, hip mobilization, knee mobilization and ankle mobilization. Each technique was applied for 3 minutes to patients.

SUMMARY:
The aim of this study was to investigate the effect of one session OMT on arterial circulation in patients with PAD.

DETAILED DESCRIPTION:
15 patients with PAD were included in the study. The OMT circulation model was applied to the participants for one session. Before and after the application, femoral artery diameter and flow rate in the patients were evaluated by doppler ultrasound

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 3 months of clinical onset of peripheral vascular disease
* Patients with ABI between 0.4-1.4
* Patients up to Stage 2b according to the Fontaine classification system

Exclusion Criteria:

* Patients undergoing vascular or endovascular surgery in the last 3 months
* Patients with unstable angina
* Patients with myocardial infarction (MI)
* Patients with stroke
* Patients with heart failure
* Patients with significant liver or renal failure (ie, dialysis)
* Acute infectious diseases
* Patients with neoplasia

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Femoral Artery Diameter Doppler Ultrasonography | 10 minutes
  Femoral artery diameter evaluated by radiologist. The femoral artery diameter unit is in mm (millimeters).
  In the evaluation, the wall contour characteristics of the vessel to be examined were evaluated and the diameter was measured. Color doppler examination was performed to determine whether the vessel contained color filling, patency, flow direction and turbulence.
  Peak systolic and end diastolic flow rates and flow pattern and flow rate were measured by spectral examination.
Femoral Artery Flow Doppler Ultrasonography | 10 minutes
  Femoral artery flow evaluated by radiologist. The femoral artery flow unit is in ml/sn (milliliter/second).
  In the evaluation, the wall contour characteristics of the vessel to be examined were evaluated and the diameter was measured. Color doppler examination was performed to determine whether the vessel contained color filling, patency, flow direction and turbulence.
  Peak systolic and end diastolic flow rates and flow pattern and flow rate were measured by spectral examination

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Ayhan ORAL, Principal Investigator — Kırıkkale University
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cerritelli F, Carinci F, Pizzolorusso G, Turi P, Renzetti C, Pizzolorusso F, Orlando F, Cozzolino V, Barlafante G. Osteopathic manipulation as a complementary treatment for the prevention of cardiac complications: 12-Months follow-up of intima media and blood pressure on a cohort affected by hypertension. J Bodyw Mov Ther. 2011 Jan;15(1):68-74. doi: 10.1016/j.jbmt.2010.03.005. Epub 2010 May 8. PMID 21147421
- [Background] Ramos-Gonzalez E, Moreno-Lorenzo C, Mataran-Penarrocha GA, Guisado-Barrilao R, Aguilar-Ferrandiz ME, Castro-Sanchez AM. Comparative study on the effectiveness of myofascial release manual therapy and physical therapy for venous insufficiency in postmenopausal women. Complement Ther Med. 2012 Oct;20(5):291-8. doi: 10.1016/j.ctim.2012.03.005. Epub 2012 May 3. PMID 22863643
- [Background] Lombardini R, Marchesi S, Collebrusco L, Vaudo G, Pasqualini L, Ciuffetti G, Brozzetti M, Lupattelli G, Mannarino E. The use of osteopathic manipulative treatment as adjuvant therapy in patients with peripheral arterial disease. Man Ther. 2009 Aug;14(4):439-43. doi: 10.1016/j.math.2008.08.002. Epub 2008 Sep 27. PMID 18824395
- [Background] Thomaz SR, Teixeira FA, de Lima ACGB, Cipriano Junior G, Formiga MF, Cahalin LP. Osteopathic manual therapy in heart failure patients: A randomized clinical trial. J Bodyw Mov Ther. 2018 Apr;22(2):293-299. doi: 10.1016/j.jbmt.2017.07.011. Epub 2017 Jul 29. PMID 29861222